CLINICAL TRIAL: NCT07286279
Title: Identifying Infertile Men Who May be Amenable to a Limited Testicular Dissection at Microdissection Testicular Sperm Extraction
Brief Title: Identifying Candidates for Limited Dissection at Microdissection TESE.
Status: Not yet recruiting | Type: Observational
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Other Study IDs: Mini incision Micro-TESE
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Non Obstructive Azoospermia; Cryptozoospermia; Oligoasthenoteratozoospermia; Male Infertility
Keywords: micro-TESE; male infertility; non-obstructive azoospermia; cryptozoospermia; oligoasthenoteratozoospermia; mini-incision
MeSH Terms: conditions — Oligospermia; Infertility, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this retrospective observational study is to learn whether certain clinical characteristics can help predict which infertile men may successfully have sperm retrieved using a less-invasive "mini-incision" version of micro-TESE. The study focuses on men with very low or absent sperm counts (non-obstructive azoospermia, cryptozoospermia, or severe OAT).

The main questions it aims to answer are:

Can sperm be successfully found using only a small, limited-dissection micro-TESE in some men?

Which clinical factors (such as hormone levels or medical history) help identify men who may benefit from this less-invasive approach?

Researchers will compare men who had successful sperm retrieval with the mini-incision alone to men who required a more extensive micro-TESE to see if certain characteristics predict which approach is likely to work.

DETAILED DESCRIPTION:
This retrospective cohort study evaluates whether preoperative clinical characteristics can help identify infertile men who are likely to achieve successful sperm retrieval through a limited-dissection, mini-incision micro-TESE. The stepwise surgical approach begins with a small equatorial incision for targeted micro-biopsies and is expanded only when sperm are not initially identified.

The study includes men who underwent their first micro-TESE at a high-volume fertility center over a 10-year period. All procedures followed a standardized surgical protocol and were performed by a single experienced surgeon, ensuring uniformity in technique.

Clinical data routinely collected before surgery, such as hormone levels, semen parameters, testicular volume, and relevant medical history, were analyzed and compared between men who required only the mini-incision and those who proceeded to an extended dissection. By examining these differences, the study aims to determine whether certain patient characteristics can predict the success with the less-invasive approach.

The findings may help guide pre-surgical counseling and support more tailored surgical planning for men with severe male factor infertility

ELIGIBILITY:
Inclusion Criteria:

* Patients with cryptozoospermia or non obstructive azoospermia that underwent a micro-TESE

Exclusion Criteria:

* Patients with a potentially reversible cause of cryptozoospermia (i.e., presence of a varicocele, febrile illness, or recent toxin exposure)
* Patients with suspected partial genital tract obstruction (i.e post-vaso-vasostomy, post-vasoepididymostomy, and low volume cryptozoospermia with ejaculatory duct obstruction)
* Patients who have previously undergone a micro-TESE, TESA or TESE procedure

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men who underwent micro-TESE procedure from March 2015 to June 2025
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Successful sperm retrieval rate defined as the presence of spermatozoa during limited dissection (mini-incision) micro-TESE | At the time of limited dissection (mini-incision)

SECONDARY OUTCOMES:
Serum FSH levels | At baseline
Serum testosterone levels | At baseline
Testicular volume | At baseline
Genetic abnormalities rate | At baseline
Procedure conversion from limited to extensive micro-TESE rate | At the time of limited dissection (mini-incision)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique ovo, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No